CLINICAL TRIAL: NCT06069349
Title: The Effect of Timing of Mobilization on Delirium in Patients After Cardiac Surgery: a Pilot Study
Brief Title: Timing of Mobilization on Delirium in Patients After Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jingyuan,Xu (Other)
Responsible Party: Sponsor-Investigator, Jingyuan,Xu, Deputy Chief Physician, Southeast University, China
Organization: Southeast University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023ZDSYLL356-P01
Record Dates: First submitted 2023-09-01; First posted 2023-10-05 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Patients After Cardiac Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual treatment (Placebo Comparator)
  Interventions: Other: usual treatment
- Early mobilization (Experimental): early mobilization in the ICU
  Interventions: Other: Early Rehabilitation

INTERVENTIONS:
Other: Early Rehabilitation — Early Rehabilitation for patients after cardiac surgery
  Arms: Early mobilization
Other: usual treatment — Patients are not allowed to exercise Early Rehabilitation
  Arms: usual treatment

SUMMARY:
Early mobilization is recommended because it is effective in improving symptoms for patients after cardiac surgery. However, the optimal timing of mobilization for postoperative patients is not unclear. How early is early? As early mobilization in the ICU is safe and may reduce healthcare costs, the goal was to assess the effect of early mobilization in the ICU on the incidence and duration of delirium.

DETAILED DESCRIPTION:
The prevalence of cardiac diseases is high, as the standard treatment for many heart diseases, a bunch of strategies are performed to improve the outcome of cardiac surgery.

Early mobilization is recommended because it is effective in improving symptoms for patients after cardiac surgery. However, the optimal timing of mobilization for postoperative patients is not unclear. How early is early? As early mobilization in the ICU is safe and may reduce healthcare costs, the goal was to assess the effect of early mobilization in the ICU on the incidence and duration of delirium.

ELIGIBILITY:
Inclusion Criteria:

* 1. > 18-year-old postoperative cardiac patient admitted to ICU, the time < 24h
* 2. Patients agree to participate in clinical research and sign informed consent before the start of the study

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for inclusion in this study:

* 1. Pregnant and lactating women
* 2. There are contraindications to getting out of bed：
* 2.1 Low cardiac output syndrome
* (1) Application of IABP or PCPS (percutaneous cardiopulmonary support)
* (2) High doses of vasoactive drugs (norepinephrine> 0.5ug/kg.min)
* (3) SBP<=80mmHg
* (4) Acrocyanosis, wet and cold
* (5) Metabolic acidosis
* (6) Urine output less than 0.5ml/kg.h for more than 2 hours
* 2.2 Heart rate greater than or equal to 120 beats per minute at rest
* 2.3 Orthostatic hypotension (systolic blood pressure less than 80 mmHg after postural change)
* 2.4 Presence of arrhythmias leading to a drop in blood pressure (e.g., decreased blood pressure due to new-onset atrial fibrillation)
* 2.5 Difficulty breathing at rest or respiratory rate greater than 30 breaths per minute
* 2.6 Postoperative bleeding (200ml in 2-3 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
duration of delirum | 7 days
  The duration of delirum in hours

SECONDARY OUTCOMES:
hospital length of stay | hospital length of stay, approximately 10 days
  hospital length of stay, approximately 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Jingyuan Xu, M.D., Study Director — Study Principal Investigator Southeast University
Locations (1):
- Zhongda hospital, Nanjing, Jiangsu, China